CLINICAL TRIAL: NCT02183142
Title: Relative Bioavailability of 7.5 mg Mobic Tablet Manufactured in China in Comparison With 7.5 mg Tablets Manufactured in Germany After a Single Oral Dose in Chinese Healthy Volunteers, Open, Randomized, Two Way Crossover Trial
Brief Title: Study of Relative Bioavailability of Mobic Manufactured in China in Comparison With Mobic Manufactured in Germany in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 107.234
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Meloxicam

ARMS (2):
- Mobic Germany (Active Comparator)
  Interventions: Drug: Mobic, China, 7.5 mg; Drug: Mobic, Germany, 7.5 mg
- Mobic China (Experimental)
  Interventions: Drug: Mobic, China, 7.5 mg; Drug: Mobic, Germany, 7.5 mg

INTERVENTIONS:
Drug: Mobic, China, 7.5 mg
Drug: Mobic, Germany, 7.5 mg

SUMMARY:
The objective of this study is to compare the pharmacokinetic parameters of the 7.5 mg Mobic tablet manufactured in china in comparison with 7.5 mg tablets manufactured in Germany

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy male volunteers as determined by result of screening
* Written informed consent in accordance with Good Clinical Practice (GCP)
* Age >= 18 and <= 40 years
* Broca > - 20% and < + 20%

Exclusion Criteria:

* Any finding of the medical examination (blood pressure, pulse rate and Electrocardiogram (ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorder
* Surgery of the gastro-intestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* Hypersensitivity to Mobic and/or non-steroidal anti-inflammatory drugs
* Intake any drugs within 1 month before randomization
* Participation in another trial with an investigational drug within the last 2 month or during the trial
* Smokers ( >= 10 cigarettes or >= 3 cigars or >= 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol or drug abuse
* Blood donation within the last 1 month
* Excessive physical activities within the last 5 days
* History of hemorrhagic diatheses
* History of gastro-intestinal ulcer, perforation or bleeding
* History of bronchial asthma

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2001-03; Primary Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax) | Up to 96 hours after drug administration
Area under the concentration-time curve of the analyte in plasma from time zero to infinity (AUC 0-infinity) | Up to 96 hours after drug administration

SECONDARY OUTCOMES:
Time to achieve Cmax (tmax) | Up to 96 hours after drug administration
Area under the concentration-time curve of the analyte in plasma from time zero to t (AUC 0-t) | Up to 96 hours after drug administration
Terminal rate constant in plasma (λ) | Up to 96 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | Up to 96 hours after drug administration
Mean residence time of the analyte (MRT) | Up to 96 hours after drug administration
Apparent clearance of the analyte in plasma following extravascular administration (CL/F) | Up to 96 hours after drug administration
Apparent volume of distribution following extravascular administration (Vd/F) | Up to 96 hours after drug administration
Number of patients with clinically relevant changes from baseline in laboratory values | Baseline, up to day 5 after last drug administration
Number of Participants with Adverse Events | Up to day 5 after last drug administration
Number of patients with clinically relevant changes from baseline in physical examination (pulse rate, systolic and diastolic blood pressure) | Baseline, up to day 5 after last drug administration
Global assessment of tolerability by investigator on a 4-point scale | Day 5 after last drug administration